CLINICAL TRIAL: NCT05911113
Title: Impact Of Sensory Re-Education Paradigm On Sensation And Quality Of Life In Patients Post-Covid 19 Polyneuropathy
Acronym: COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Younes Ali Khadour, principle investigator younes ali khadour, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004416
Record Dates: First submitted 2023-06-17; First posted 2023-06-20 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Post-COVID-19 Syndrome
Keywords: post-covid 19 polyneuropathy; sensory re-education paradigm; sensation; quality of life
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: sensory re-education and traditional therapy
Who Masked: Participant, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sensory re-education training (Experimental): the patients will receive sensory re-education training three times a week for six weeks
  Interventions: Other: sensory re-education training; Other: traditional treatment
- traditional treatment (Active Comparator): the patients will receive traditional treatment three times a week for six weeks
  Interventions: Other: traditional treatment

INTERVENTIONS:
Other: sensory re-education training — the patients will receive sensory re-education training in the form of texture discrimination training, limb position sense and tactile object recognition
  Arms: sensory re-education training
Other: traditional treatment — the Patients in this group will receive traditional treatment in the form of proprioception neuromuscular facilitation (PNF) and graduated active and resisted wrist and hand muscle strengthening exercises.

SUMMARY:
This study will be conducted to investigate the effect of a sensory re-education paradigm on sensation and proprioception in patients with post covid-19 neuropathy.

DETAILED DESCRIPTION:
The Coronavirus disease has profoundly impacted the world, altering the functioning of the population and health system. it is so far affected more than 532 million cases and 6.3 million confirmed deaths (WHO., 2020). Recent studies documented that COVID-19-associated peripheral neuropathy is a common and frequent problem, with neuro-muscular complications. This phenomenon is widespread in those with comorbidities, such as diabetes mellitus, which may result from immune processes or as side effects of some medications used to manage COVID-19 symptoms, such as hydroxychloroquine, clindamycin, and steroids. To a lesser extent, prolonged hospitalization may cause entrapment neuropathy (peripheral nerve compression). Most physiotherapists focus on motor improvements rather than sensibility improvements though the sensory system may have the upper hand in improving motor function. Therefore; the sensory re-education paradigm should be assessed in randomized trials with a blinded assessment of functional outcomes to evaluate its effectiveness in patients with post covid-19 neuropathic patients. Currently, there is not enough research addressing the impact of the sensory re-education paradigm on sensation and quality of life in neuropathic patients post-covid19. forty patients will be assigned randomly into two equal groups; the study group will receive sensory re-education paradigm and traditional treatment while the control group will receive traditional treatment only.

ELIGIBILITY:
Inclusion Criteria:

Patients from both genders (male and female). The age of participants ranged from 30 to 40 years old. Participants were required to live in Egypt during the pre-covid and COVID-19 pandemic.

Patients with confirmation of previous covid19 infection PCR TEST. Patients meeting the guide line of world health organization (WHO) of long/post-covid 19 syndromes.

Patients with unknown prior neuropathy. Patients with neuropathy confirmed by EDX with a sensory nerve conduction velocity.

Exclusion Criteria:

Patients with Diabetes mellitus (DM), Rheumatology and Guillain-Barré syndrome (GBS).

Infection other than covid19 leading to sensory neuropathy. Traumatic or compressive lesions leading to central nervous system (CNS), peripheral nervous system (PNS) damages.

Previous surgeries or medications leading to neuropathy.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
disability of life | up to six weeks
  disability of life will be measured using the Arabic, validated version of WHOQOL-BREF questionnaire. The scale consists of 26 items; the first two items address an individual's perception of his/her overall quality of life and health, respectively, and the remaining 24 items assess the four quality of life domains; Physical Health (seven items), Psychological (six items), Social Relationships (three items), and Environment (eight items). Each item is rated on a five-point Likert scale. The final scores were converted into a linear scale between 0 and 100 according to the scoring guidelines where higher scores indicate higher disability.

SECONDARY OUTCOMES:
Tactile sensation | up to six weeks
  The Semmes Weinstein Monofilament (SWM) tool will be used to assess cutaneous sensibility threshold. This is to assess touch detection thresholds of the hand and fingers. The short version (pocket filaments) with five filaments from 0.07 to 300 g was used. The touch detection thresholds were scored on a 0 to 5-point scale, where 5 represents the thinnest filament and 0 represents the largest filament. Three different positions of the hand were tested: the fingertip of fingers, proximal phalanx of fingers, and palm of the hand yielding a total sum score of 15 points
hand grip strength | up to six weeks
  The hand-held dynamometer will be used to assess hand grip strength
joint position error | up to six weeks
  The laser-pointer assisted angle reproduction test will be used to assess the joint position error of wrist joint.The test person will be sitting on a hand-rested chair the wrist will be free out of the hand-rest of the chair, the chair is seated at a marked line on the floor that being drawn parallelly and in one-meter distance to a target board fixed on the opposite wall. A pointing laser will be fixed at the dorsum of the hand. The test person will be asked to raise their affected wrist from neutral position to aim for assigned points at 10°, 30° and 45°. The neutral position is defined as arbitrary zero. Values at a positive angels represent flexion angels. The negative angels will represent extension angels. The patient is required to memorize the different joint positions. In the next step, the patient's eyes were covered to inhibit visual control. Then they were asked to reproduce the same joint positions as before in a randomized order.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt